CLINICAL TRIAL: NCT01460199
Title: A Multi Center, Double-Blind, Two-Arm,Placebo Controlled, Randomized Safety and Tolerability Study of CTP-499 in Non-Dialysis Patients With Stage 3 Chronic Kidney Disease
Brief Title: Safety & Tolerability Study of CTP-499 in Patients With Moderate Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP505.1003
Record Dates: First submitted 2011-10-20; First posted 2011-10-26 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Stage 3 Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — 1-(5-hydroxyhexyl)-3,7-dimethylxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: placebo
- CTP-499 (Experimental)
  Interventions: Drug: CTP-499

INTERVENTIONS:
Drug: CTP-499 — 3 X 200 mg tablets (QD for 2 weeks)
  3 x 200 mg tablets (BID for 2 weeks)
  Arms: CTP-499
Drug: placebo — tablets
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of treatment with CTP-499 in non-dialysis patients associated with moderate chronic kidney disease.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of treatment with CTP-499 starting with 600 milligrams (mg) once a day (QD) for 2 weeks followed by 600 mg twice a day (BID) for 2 weeks in non-dialysis patients associated with moderate chronic kidney disease defined as an estimated Glomerular Filtration Rate or eGFR that is 30-59 mL/min/1.73m2

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of chronic kidney disease
* If taking antihypertensive and antidiabetes medications, regimen must be stable for a minimum of 4 weeks
* Patient has systolic blood pressure less than or equal to 160 mm Hg and diastolic blood pressure less than or equal to 95 mm Hg

Exclusion Criteria:

* Patient has concurrent condition such as uncontrolled inflammatory disease, acute infection or clinically unstable autoimmune, endocrine, neurological, psychiatric, retinal, cardiovascular, bronchopulmonary, hepatic, gastrointestinal or musculoskeletal disorder
* Patient has acute, active and/or current unstable renal impairment disease
* Patient has been hospitalized for acute renal failure in the past year
* Patient has active malignancy or a history of neoplastic disease
* Patient has QTc interval > 450 milliseconds
* Patient is currently on cytotoxic or other immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety measures | 4 weeks
  number of adverse events, vital signs, ECGs, clinical laboratory measures and physical exams

SECONDARY OUTCOMES:
Pharmacokinetic Profile | 4 weeks
  Time Frame: Predose, 0, 1, 2, 3, 4, 6, 8, 12, 18, 24 hours Cmax, Tmax, Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: James Shipley, MD, Study Director — Concert Pharmaceuticals
Locations (3):
- United States (3):
  - West Coast Clinical Trials, Costa Mesa, California
  - Southern California Clinical Research, Garden Grove, California
  - Orange County Research Center, Tustin, California